CLINICAL TRIAL: NCT01102127
Title: Accuracy of Ultrasound Elastastography in Thyroid Nodular Disease.
Brief Title: Elastography in Thyroid Nodules
Status: Completed | Type: Observational
Sponsor: Castilla-León Health Service (Other)
Responsible Party: Alfonso Vidal-Casariego, Complejo Asistencial de León
Other Study IDs: TNUS122009
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-04

CONDITIONS: Nodular Goiter; Thyroid Cancer
Keywords: elastography; thyroid nodule; fine-needle aspiration
MeSH Terms: conditions — Goiter, Nodular; Thyroid Neoplasms; Thyroid Nodule | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Thyroid cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Goiter: Patients with nodular goiter
  Interventions: Device: Elastography

INTERVENTIONS:
Device: Elastography — Performance of US, elastography and FNA.

SUMMARY:
Nodular goiter is a highly prevalent disease in iodine-deficient areas. Usually nodule assessment includes ultrasonography (US) and fine-needle aspiration (FNA), but some benign nodules can hardly be distinguished from carcinomas. Elastography measures tissue elasticity using sonography, as malignancy is related to stiffness of solid organs. The investigators have designed a study to evaluate the diagnostic accuracy of elastography in nodular goiter. Consecutive patients will be assessed using US, FNA and elastography; the latter will be compared with cytology. Specificity, sensitivity, and predictive values will be calculated.

DETAILED DESCRIPTION:
Aims:

Primary aim: to evaluate the diagnostic accuracy of elastography in thyroid nodules from a low-risk of thyroid cancer population.

Secondary aim: to evaluate the usefulness of elastography to detect carcinomas in thyroid nodules with indeterminate FNA.

Patient selection:

Inclusion criteria:

* Age > 18 yr.
* Recruitment in Endocrinology Clinics.
* Nodular goiter.
* Multinodular goiter with dominant nodule > 1 cm.

Exclusion criteria:

* Toxic nodules
* Non-accessible nodules to US or FNA
* Cystic nodules
* Nodules with calcifications in egg rind
* Contraindication for FNA

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yr.
* Recruitment in Endocrinology surgery.
* Nodular goiter.
* Multinodular goiter with dominant nodule > 1 cm.

Exclusion Criteria:

* Toxic nodules
* Non-accessible nodules to US or FNA
* Cystic nodules
* Nodules with calcifications in egg rind
* Contraindication of FNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population with nodular goiter.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of elastography for thyroid cancer | 1 day
  Sensitivity, specifity, predictive values

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Vidal-Casariego, MD, Principal Investigator — Complejo Asistencial de León
Locations (1):
- Complejo Asistencial de León, León, León, Spain

REFERENCES:
- [Background] Dighe M, Kim J, Luo S, Kim Y. Utility of the ultrasound elastographic systolic thyroid stiffness index in reducing fine-needle aspirations. J Ultrasound Med. 2010 Apr;29(4):565-74. doi: 10.7863/jum.2010.29.4.565. PMID 20375375
- [Background] Tonacchera M, Pinchera A, Vitti P. Assessment of nodular goitre. Best Pract Res Clin Endocrinol Metab. 2010 Feb;24(1):51-61. doi: 10.1016/j.beem.2009.08.008. PMID 20172470
- [Background] Luo S, Kim EH, Dighe M, Kim Y. Screening of thyroid nodules by ultrasound elastography using diastolic strain variation. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:4420-3. doi: 10.1109/IEMBS.2009.5332744. PMID 19963828
- [Background] Friedrich-Rust M, Sperber A, Holzer K, Diener J, Grunwald F, Badenhoop K, Weber S, Kriener S, Herrmann E, Bechstein WO, Zeuzem S, Bojunga J. Real-time elastography and contrast-enhanced ultrasound for the assessment of thyroid nodules. Exp Clin Endocrinol Diabetes. 2010 Oct;118(9):602-9. doi: 10.1055/s-0029-1237701. Epub 2009 Oct 23. PMID 19856256
- [Derived] Vidal-Casariego A, Lopez-Gonzalez L, Jimenez-Perez A, Ballesteros-Pomar MD, Kyriakos G, Urioste-Fondo A, Alvarez-San Martin R, Cano-Rodriguez I, Jimenez-Garcia de la Marina JM. Accuracy of ultrasound elastography in the diagnosis of thyroid cancer in a low-risk population. Exp Clin Endocrinol Diabetes. 2012 Nov;120(10):635-8. doi: 10.1055/s-0032-1323804. Epub 2012 Oct 16. PMID 23073921